CLINICAL TRIAL: NCT04362735
Title: Efficacy of Vedolizumab in Crohn's Disease Patients Naive to Biological Therapy: a Brazilian Multicentric Observational Real-world Study
Brief Title: Efficacy of Vedolizumab in Crohn's Disease Patients Naive to Biological Therapy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Pontifícia Universidade Católica do Paraná (Other)
Collaborators: Takeda (Industry)
Responsible Party: Principal Investigator, Roberto Pecoits-Filho, Professor, Pontifícia Universidade Católica do Paraná
Other Study IDs: IISR-2020-103104
Record Dates: First submitted 2020-04-19; First posted 2020-04-27 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Crohn Disease
Keywords: vedolizumab
MeSH Terms: conditions — Crohn Disease | interventions — vedolizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study group: All patients using vedolizumab for Crohn's disease as first biologic agent (all patients naive to previous biological therapy)
  Interventions: Drug: Vedolizumab

INTERVENTIONS:
Drug: Vedolizumab — Vedolizumab 300 mg at weeks 0, 2 and 6 as induction. Maintenance every 4 or 8 weeks, as on-label recommendations.

SUMMARY:
INTRODUCTION: Vedolizumab is a gut selective anti-integrin agent which binds to the alfa4beta7 integrin, preventing its coupling to the endothelial MadCAM-1. It reduces leucocyte trafficking from the endothelium consequently reducing intestinal tissue inflammation. There is scarce evidence on the use of vedolizumab in CD in Brazil, mostly in patients with no previous biological therapy, where the drug seems to have a more adequate therapeutic potential.

Tha primary aim of the study is to analyze clinical remission rates at weeks 12, 26 and 52, and at last follow-up on naive CD patients submitted to vedolizumab therapy. Secondary outcomes will be clinical response rates at weeks 12, 26 and 52, and at last follow-up; endoscopic remission rates in colonoscopies performed; persistence of drug therapy over time; adverse events during treatment with vedolizumab and rates of abdominal surgery during therapy.

METHODS: A retrospective, longitudinal, observational study will be performed with patients with CD who used Vedolizumab at any time of their treatment as the first biologic option, after failure of conventional therapy. Following the induction dose of 300 mg at weeks 0, 2 and 6, and maintenance of 300 mg every 8 weeks, patients will be followed up to 52 weeks (1 year) or more (last follow-up captured). Records of the clinical evaluations at week 12, 26 and 52, and last follow-up, will be checked according to the HBI and PGA to define clinical response or clinical remission. Colonoscopies will also be checked to evaluate mucosal healing. Electronic charts will be reviewed also to analyze adverse events and surgery during therapy.

DETAILED DESCRIPTION:
INTRODUCTION: Inflammatory bowel diseases (IBD) are a group of chronic, idiopathic and immune-mediated diseases, mainly represented by Crohn's disease (CD) and Ulcerative Colitis (UC). There is a broad therapeutic spectrum according to the degree of disease activity, extension and behavior, from aminosalicylates to biological therapy. Tumor necrosis factor (TNF) alpha inhibitors were the first class of biological therapy approved for IBD. However, some patients do not respond to treatment (primary non-responders) or lose response over time (secondary loss of response). With a different mechanism of action, the class of anti-integrin monoclonal antibodies, represented by natalizumab and vedolizumab, has recently expanded. Vedolizumab is a gut selective anti-integrin that binds to the alfa4beta7 integrin, preventing its coupling to the endothelial MadCAM-1. In this way, it reduces the process of lymphocyte migration and reduces intestinal tissue inflammation. Multicentric real life studies with vedolizumab in UC and CD showed the efficacy and safety of the drug. More recently, a head-to-head trial comparing the efficacy of vedolizumab against adalimumab in UC demonstrated superiority of vedolizumab in comparison to the subcutaneous anti-TNF agent, defining positioning of the drug as an adequate first option in therapeutic sequencing. There is no head to head trial comparing vedolizumab against other agents in CD. Indeed, there is a lack of studies on the use of vedolizumab in CD in Brazil, mostly in biologic naïve patients, where the drug seems to have a more adequate therapeutic potential.

OBJECTIVES:

1. Primary objective: to analyze clinical remission rates [defined as a Harvey-Bradshaw index (HBI) of equal or lower than 4 for Crohn's disease (CD)] at weeks 12, 26 and 52, and at last follow-up.
2. Secondary objectives: to analyze clinical response rates (defined as a reduction at the HBI of equal or more than 3 points for CD and according to physician global assessment - PGA) at weeks 12, 26 and 52, and at last follow-up; to analyze endoscopic remission rates (defined as absence of ulcers in CD) in colonoscopies performed; to analyze persistence of drug therapy over time; to analyze adverse events during treatment with vedolizumab and rates of abdominal surgery during therapy.

METHODS: This project is already approved by the Institutional Review Board (IRB) from the Catholic University of Paraná, Brasil. A retrospective, longitudinal, observational study will be performed with patients with CD who used Vedolizumab at any time of their treatment as the first biologic option, after failure of conventional therapy. Inclusion criteria: Patients with CD, who used vedolizumab as the first biological agent during medical treatment, after failure of conventional therapy (aminosalicylates, steroids and/or immunomodulators such as azathioprine and methotrexate). Exclusion criteria: Patients with UC, other causes of intestinal inflammation (ischemic or infectious colitis, for example) non-IBD related, IBD-undetermined not defined as CD or UC will be excluded from the analysis. Patients with vedolizumab who had previous exposure to anti-TNF agents will also be excluded. Pregnant and pediatric patients (less than 18 years old) will also be excluded. Following the induction dose of 300 mg at weeks 0, 2 and 6, and maintenance of 300 mg every 8 weeks, patients will be followed up to 52 weeks (1 year) or more (last follow-up captured). Records of the clinical evaluations at week 12, 26 and 52, and last follow-up, will be checked according to the HBI for CD, and PGA to define clinical response or clinical remission. Colonoscopies will also be checked to evaluate mucosal healing.

ELIGIBILITY:
Inclusion Criteria:

- Patients with CD (any location)who used vedolizumab as the first biological agent during medical treatment, after failure of conventional therapy (5-ASA, steroids and/or immunomodulators such as azathioprine and methotrexate).

Exclusion Criteria:

* Patients with UC
* Patients with other causes of intestinal inflammation (ischemic or infectious colitis, for example) non-IBD related
* Patients with IBD-undetermined not defined as CD or UC
* Patients with vedolizumab who had previous exposure to anti-TNF agents
* Pregnant patients
* Pediatric patients (less than 18 years old)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients using vedolizumab as first option of biological therapy for CD of any location.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2021-01-20 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
Clinical remission | 12 weeks
  HBI index ≤ 4
Clinical remission | 26 weeks
  HBI index ≤ 4
Clinical remission | 52 weeks
  HBI index ≤ 4

SECONDARY OUTCOMES:
Clinical response | 12 weeks
  reduction in HBI index ≥ 3 points + PGA
Clinical response | 26 weeks
  reduction in HBI index ≥ 3 points + PGA
Clinical response | 52 weeks
  reduction in HBI index ≥ 3 points + PGA
Mucosal healing | through study completion, an average of 52 weeks
  absence of ulcers at colonoscopy
Need for major surgery during treatment | through study completion, an average of 52 weeks
  Any major abdominal surgery during therapy with vedolizumab

CONTACTS AND LOCATIONS:
Overall Officials: Paulo Kotze, phd, Principal Investigator — Professor of postgraduate program

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Perin RL, Damiao AOMC, Flores C, Ludvig JC, Magro DO, Miranda EF, Moraes AC, Nones RB, Teixeira FV, Zeroncio M, Kotze PG. VEDOLIZUMAB IN THE MANAGEMENT OF INFLAMMATORY BOWEL DISEASES: A BRAZILIAN OBSERVATIONAL MULTICENTRIC STUDY. Arq Gastroenterol. 2019 Sep 30;56(3):312-317. doi: 10.1590/S0004-2803.201900000-58. eCollection 2019. PMID 31633731
- [Result] Kopylov U, Verstockt B, Biedermann L, Sebastian S, Pugliese D, Sonnenberg E, Steinhagen P, Arebi N, Ron Y, Kucharzik T, Roblin X, Ungar B, Shitrit AB, Ardizzone S, Molander P, Coletta M, Peyrin-Biroulet L, Bossuyt P, Avni-Biron I, Tsoukali E, Allocca M, Katsanos K, Raine T, Sipponen T, Fiorino G, Ben-Horin S, Eliakim R, Armuzzi A, Siegmund B, Baumgart DC, Kamperidis N, Maharshak N, Maaser C, Mantzaris G, Yanai H, Christodoulou DK, Dotan I, Ferrante M. Effectiveness and Safety of Vedolizumab in Anti-TNF-Naive Patients With Inflammatory Bowel Disease-A Multicenter Retrospective European Study. Inflamm Bowel Dis. 2018 Oct 12;24(11):2442-2451. doi: 10.1093/ibd/izy155. PMID 29788318
- [Result] Schreiber S, Dignass A, Peyrin-Biroulet L, Hather G, Demuth D, Mosli M, Curtis R, Khalid JM, Loftus EV Jr. Systematic review with meta-analysis: real-world effectiveness and safety of vedolizumab in patients with inflammatory bowel disease. J Gastroenterol. 2018 Sep;53(9):1048-1064. doi: 10.1007/s00535-018-1480-0. Epub 2018 Jun 4. PMID 29869016